CLINICAL TRIAL: NCT06048133
Title: Study of Gemcitabine, Cisplatin, Quemliclustat (AB680) and Zimberelimab (AB122) During First-line Treatment of Advanced Biliary Tract Cancers (QUIC)
Brief Title: Study of Gemcitabine, Cisplatin, AB680 and AB122 During First Line Treatment of Advanced Biliary Tract Cancers (QUIC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nataliya Uboha (Other)
Collaborators: Arcus Biosciences, Inc. (Industry); Gilead Sciences (Industry); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor-Investigator, Nataliya Uboha, Sponsor Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-GI22-564
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Carcinoma; Cholangiocarcinoma; Bile Duct Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Gemcitabine; Cisplatin; zimberelimab; quemliclustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Quemliclustat (AB680), zimberelimab (AB122), gemcitabine, and cisplatin in subjects with untreated advanced BTC. Quemliclustat IV: Day 1, 15, and 29 of each cycle; Zimberelimab IV: Day 1 and 22 of each cycle; Gemcitabine IV: Day 1, 8, 22 and 29 of each cycle; Cisplatin IV: Day 1, 8, 22 and 29 of Cycles 1-4 only.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Zimberelimab; Drug: Quemliclustat

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine IV: Day 1, 8, 22, and 29 every 42 days
Drug: Cisplatin — Cisplatin IV: Day 1, 8, 22, and 29 every 42 days of Cycles 1-4 only.
Drug: Zimberelimab — Zimberelimab IV: Day 1 and 22 every 42 days
  Other Names: AB122
Drug: Quemliclustat — Quemliclustat IV: Day 1, 15, 29 every 42 days
  Other Names: AB680

SUMMARY:
This is a phase 2 study of gemcitabine, cisplatin, zimberelimab (AB122) and quemliclustat (AB680) in subjects with untreated advanced biliary tract cancers (BTC). The study will include a safety run-in involving 6 study participants. The goal of the safety run-in is to screen for early safety signals of the proposed drug combination. Trial enrollment can continue while full safety assessment is being completed for the first 6 subjects.

Participants will receive 4 cycles of combination therapy as described. After 4 cycles (~6 months), cisplatin will be discontinued, while gemcitabine, zimberelimab (AB122), and quemliclustat (AB680) will be continued. Subjects will be treated until disease progression or development of intolerable toxicities. In total, there will be up to 39 participants on the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cytologically or histologically confirmed BTC by AJCC version 8.
2. Patients must have late stage (locally advanced, recurrent or metastatic) BTC. Patients must not have received systemic treatment for advanced disease. Prior adjuvant therapy is allowed as long as recurrences occurred 6 months or later from all treatment completion.
3. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
4. Age ≥ 18 years at the time of consent.
5. ECOG Performance Status of 0-2 within 28 days prior to registration.
6. Presence of measurable or evaluable disease, as defined by RECIST v1.1.
7. Adequate organ function as detailed in the protocol.
8. Females of childbearing potential who are sexually active with a male able to father a child must have a negative pregnancy test (serum or urine) within 14 days prior to registration. NOTE: Biliary cancer may secrete hormones to produce a false-positive pregnancy test. Female subjects of childbearing potential with a positive pregnancy test should have a thorough history and additional work up as determined by the treating physician to rule out pregnancy (e.g. serial βHCG measurements, ultrasound). Once pregnancy has been ruled out, the subject may proceed with screening and enrollment.
9. Females of childbearing potential who are sexually active with a male able to father a child must be willing to abstain from heterosexual vaginal intercourse or use an effective method(s) of contraception from the time of informed consent, during the study and for up to 14 months after the last dose of study drug(s). Males able to father a child must be willing to abstain from heterosexual vaginal intercourse or to use an effective method(s) of contraception from initiation of treatment, during the study and for up to 11 months after the last dose of study drug(s). See the protocol for specific timeframes for each drug.
10. Ability of the subject to understand and comply with study procedures for the entire length of the study, as determined by the enrolling physician or protocol designee.

Exclusion Criteria:

1. Prior therapy with gemcitabine, cisplatin, or any immune checkpoint inhibitors for the treatment of BTC.
2. Known hypersensitivity to recombinant proteins, or any excipient contained in treatment medication formulations.
3. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

   NOTE: participants with asthma who require intermittent use of bronchodilators, inhaled corticosteroids, or local corticosteroid injections will not be excluded from this study.
4. History of solid organ or allogeneic bone marrow transplantation.
5. Pregnant or breastfeeding. NOTE: breast milk cannot be stored for future use while the mother is being treated on study.
6. Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are not eligible for this trial.
7. Untreated central nervous system (CNS) metastasis. Screening of asymptomatic patients for CNS metastasis is not required for enrollment.
8. Underlying medical conditions that, in the Investigator's or Sponsor's opinion, will make the administration of IP(s) hazardous, including but not limited to

   * Interstitial lung disease, including history of interstitial lung disease or non-infectious pneumonitis.
   * Active viral, bacterial, or fungal infections requiring parenteral treatment within 14 days of the initiation of the study treatments.
9. History of trauma or major surgery within 28 days prior to the first dose of IP. (Note that placement of central venous access catheter (e.g., port or similar) is not considered a major surgical procedure.
10. Treatment with palliative radiation therapy within 14 days of study treatment initiation.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Significant dementia or other mental condition that precludes the participant's ability to consent to the study.
13. Use of any live vaccines against infectious diseases within 4 weeks (28 days) of initiation of investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Estimate the progression free survival (PFS) with gemcitabine, cisplatin, quemliclustat (AB680) and zimberelimab (AB122) in patients with advanced BTCs. | 2 years
  Progression free survival (PFS), as determined by RECIST v1.1, is defined as the time from study registration to the date of documented disease progression or death from any cause.

SECONDARY OUTCOMES:
Estimate the overall survival (OS) | 2 years
  Overall survival, defined as the time from study enrollment to date of death due to any cause. Subjects without documented death at the time of analysis will be censored at the date of last known contact.
Estimate the objective response rate (ORR) | 2 years
  Objective response rate, defined as the proportion of subjects with a complete or partial response to treatment according to RECIST, version 1.1.
Estimate the disease control rate (DCR) | 2 years
  Disease control rate, defined as the proportion of subjects with stable disease, complete or partial response to treatment according to RECIST, version 1.1.
Estimate the duration of response (DOR) | 2 years
  Duration of Response (DOR) is defined as the time that measurement criteria are met for complete or partial response according to RECIST 1.1 (whichever status is recorded first) until the date recurrent or progressive disease, or death, is objectively documented (taking as reference for progressive disease the smallest measurements recorded since treatment started).
Evaluate safety of the proposed drug combination. | 2 years
  Safety and tolerability will be assessed by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Nataliya Uboha, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Wisconsin, Madison, Wisconsin